CLINICAL TRIAL: NCT00188383
Title: Effects of NMDA-Receptor Antagonism on Hyperalgesia, Opioid Use, and Pain After Radical Prostatectomy in Young and Elderly Patients
Brief Title: Effects of N-Methyl-D-Aspartate (NMDA)-Receptor Antagonism on Hyperalgesia, Opioid Use, and Pain After Radical Prostatectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 94759-200109MCT
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2005-09

CONDITIONS: Hyperalgesia; Pain; Prostate Cancer
Keywords: Hyperalgesia; Quantitative Sensory Testing; Pain; Opioid use; Elderly
MeSH Terms: conditions — Hyperalgesia; Pain; Prostatic Neoplasms | interventions — Amantadine

INTERVENTIONS:
Drug: Amantadine

SUMMARY:
The primary aim is to determine whether perioperative NMDA-receptor antagonism has differential effects on postoperative pain, hyperalgesia and morbidity in younger and older patients. In order to achieve this aim, the researchers propose to conduct the first randomized, double-blind placebo-controlled study designed to investigate age differences in the effects of perioperative oral administration of an NMDA-receptor antagonist (amantadine) in men undergoing radical prostatectomy. In addition, age differences in psychosocial factors and the pharmacological properties of amantadine and morphine will be measured to control for, and clarify, their contribution to the differences found.

The specific objectives of the study are to:

1. investigate the effects of perioperative NMDA receptor blockade on postoperative hyperalgesia, pain and analgesic consumption in young and elderly men
2. assess age differences in the intensity and course of secondary hyperalgesia after surgery

DETAILED DESCRIPTION:
The immediate postoperative period is associated with spontaneous pain and hyperalgesia, i.e., increased pain response (both intensity and duration) to normally painful stimuli following tissue injury or damage.

The development and maintenance of secondary hyperalgesia depend on complex plastic changes in spinal cord dorsal horn cells after peripheral injury or damage. Afferent impulses signaling the damage are carried to the dorsal horn by slowly conducting, unmyelinated C-fibres. C-fibres release glutamate which acts at three receptor types: metabotropic, kainate/AMPA and NMDA. NMDA receptor activation, through a complex cascade of intracellular events, results in dorsal horn neuron hyperexcitability or central sensitization. These cells have increased spontaneous activity, decreased threshold, increased response to afferent input, prolonged afterdischarge to repeated stimulation, and an expansion of receptive fields. Central sensitization is expressed behaviorally as secondary hyperalgesia and contributes to prolonged postoperative pain. It also may trigger pathological reorganization of neural circuitry leading to the development of chronic postsurgical pain. Through these processes, tissue injury may have profound effects on the CNS that long outlast the injury.

In animal models of pain, NMDA agonists induce central sensitization and hyperalgesia whereas antagonists decrease or prevent hyperalgesia. In humans, NMDA-receptor antagonism decreases secondary hyperalgesia subsequent to experimentally-induced pain.

Perioperative administration of NMDA antagonists, that is, before, during and after surgery, may be the ideal intervention to block the initiation and maintenance of central sensitization. Several studies have found that this intervention reduces postoperative hyperalgesia, pain, and analgesic use; however, others have not found these effects. This is not surprising given the variability across studies in factors such as surgical procedure, extent and nature of tissue damage, duration of surgery, pharmacokinetics of the agent(s) tested, and intraoperative and postoperative analgesia. Nonetheless, the weight of the evidence suggests that preventing or minimizing central sensitization reduces pain and analgesic requirements.

Co-administration of NMDA antagonists and opioids has been advocated as an effective approach. The combination of morphine and amantadine should reduce postoperative pain by inducing analgesia through actions on opioid-mediated receptor systems and by reducing hyperalgesia via NMDA receptor-mediated events . The combination also should produce fewer opioid-related adverse effects due to the anticipated opioid-sparing effect. The present proposal describes the first direct comparison of perioperative NMDA receptor blockade coupled with intra- and post-operative opioid administration in young and elderly patients. In order to minimize the influence of other perioperative factors on the outcome variables, all patients will undergo the same surgical procedure and anesthetic protocol. Furthermore, factors that cannot readily be standardized (e.g., surgical duration, mood) will be measured and controlled for statistically. This increases the internal validity of the proposed study and our ability to detect age and drug effects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and write English;
2. Age 18-59 or >= 60 years;
3. American Society of Anesthesiologists Class 1 to 3;
4. Scheduled for elective radical prostatectomy;
5. Body weight between 50-110 kg, body mass index (BMI) <= 30.

Exclusion Criteria:

1. Significant central nervous system (CNS), respiratory, cardiac, hepatic, renal or endocrine dysfunction and/or any significant sequelae;
2. Contraindications, allergies to, and/or past adverse reactions to opioid analgesics, amantadine or nonsteroidal anti-inflammatory drugs (NSAIDS);
3. Current Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) Axis I disorder or cognitive dysfunction or history of this within the last year;
4. History of epilepsy or other seizures;
5. History of chronic pain of at least 6 months duration;
6. History of long term opioid use for chronic pain of at least 6 months duration;
7. History of long term use of amantadine or other antiparkinsonian drug;
8. Ingestion of antitussive medication (dextromethorphan) within the 48 hours before surgery;
9. History of alcohol or drug dependency/abuse of at least 6 months duration

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2004-01; Study Completion 2006-12

PRIMARY OUTCOMES:
To investigate the effects of perioperative NMDA receptor blockade on postoperative hyperalgesia, pain and analgesic consumption in young and elderly men

SECONDARY OUTCOMES:
To assess age differences in the intensity and course of secondary hyperalgesia after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Gagliese, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada